CLINICAL TRIAL: NCT01912937
Title: ProspectIve, SingLe-Arm, MuLti-Center, Pharmacokinetic Study to EvalUate TreatMent of Obstructive SupErficial Femoral Artery or Popliteal LesioNs With A Novel PacliTaxel-CoatEd Percutaneous Angioplasty Balloon
Brief Title: Pharmacokinetic Study of Drug-coated Angioplasty Balloons in the Superficial Femoral or Popliteal Arteries:
Acronym: PK
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Spectranetics Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TP-1363
Record Dates: First submitted 2013-07-10; First posted 2013-07-31 (Estimated); Last update posted 2017-10-18 (Actual); Status verified 2017-10

CONDITIONS: Peripheral Artery Disease
Keywords: Paclitaxel; Percutaneous Transluminal Angioplasty; Balloon Catheter; Pharmacokinetic; Peripheral Artery Disease; PAD
MeSH Terms: conditions — Peripheral Arterial Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- DCB Arm (Experimental): Angioplasty treatment with the CVI Paclitaxel-Coated, Percutaneous Transluminal Angioplasty (PTA) Balloon Catheter (CVI Paclitaxel-coated PTA Catheter)
  Interventions: Device: Angioplasty treatment with the CVI Drug-coated Balloon (DCB)

INTERVENTIONS:
Device: Angioplasty treatment with the CVI Drug-coated Balloon (DCB) — Angioplasty treatment with the CVI Paclitaxel-Coated, Percutaneous Transluminal Angioplasty (PTA) Balloon Catheter (CVI Paclitaxel-coated PTA Catheter)

SUMMARY:
To describe the pharmacokinetics of paclitaxel in the blood delivered from a paclitaxel coated percutaneous angioplasty balloon catheter as a result of treatment of de novo or restenotic lesion(s), occluded/stenotic or re-occluded/restenotic lesion(s).

DETAILED DESCRIPTION:
This study investigates the inhibition of restenosis using the CVI Paclitaxel-coated PTA Catheter in the treatment of de-novo occluded/stenotic or re-occluded/ restenotic superficial femoral or popliteal arteries. The proposed clinical study will be a prospective, non-randomized, single arm, multi-center, pharmacokinetic study. The objective of the study is to describe the pharmacokinetics of paclitaxel in the blood delivered from the CVI Paclitaxel-coated PTA Catheter as a result of de novo occluded/restenotic or re-occluded/restenotic lesion(s).

ELIGIBILITY:
Inclusion Criteria:

* Male or non-pregnant female greater than or equal to 18 years of age.
* Subjects with symptomatic leg ischemia, requiring treatment of the Superficial Femoral Artery (SFA) or popliteal artery.

Exclusion Criteria:

* Pregnant or lactating females.
* Known intolerance to study medications, paclitaxel or contrast agents that in the opinion of the investigator cannot be adequately pre-treated.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2013-06 (Actual); Primary Completion 2016-06 (Actual); Study Completion 2017-07 (Actual)

PRIMARY OUTCOMES:
Paclitaxel Levels | up to 6 months
  Measurement of paclitaxel concentration in the circulating blood immediately after last balloon deployment, 1, 4, 24 hours, 7, 14, 30, 60 days and 6 months (if applicable) post-procedure.
Freedom from Events as a Safety Measure (Composite) | up to 12 months
  Freedom from device and procedure-related death through 30 days post-procedure; and freedom from target limb major amputation and clinically-driven target lesion revascularization through 12 months post-procedure.

SECONDARY OUTCOMES:
Measurements of Pharmacokinetics variables: Cmax, Tmax, AUC | (0-t) and half-life

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Holden, MD, Principal Investigator — Auckland City Hospital
Locations (2):
- New Zealand (2):
  - Auckland City Hospital, Auckland
  - Clinical Trials New Zealand, Hamilton

REFERENCES:
- [Derived] Gray WA, Jaff MR, Parikh SA, Ansel GM, Brodmann M, Krishnan P, Razavi MK, Vermassen F, Zeller T, White R, Ouriel K, Adelman MA, Lyden SP. Mortality Assessment of Paclitaxel-Coated Balloons: Patient-Level Meta-Analysis of the ILLUMENATE Clinical Program at 3 Years. Circulation. 2019 Oct;140(14):1145-1155. doi: 10.1161/CIRCULATIONAHA.119.040518. Epub 2019 Sep 30. PMID 31567024
- [Derived] Krishnan P, Faries P, Niazi K, Jain A, Sachar R, Bachinsky WB, Cardenas J, Werner M, Brodmann M, Mustapha JA, Mena-Hurtado C, Jaff MR, Holden AH, Lyden SP. Stellarex Drug-Coated Balloon for Treatment of Femoropopliteal Disease: Twelve-Month Outcomes From the Randomized ILLUMENATE Pivotal and Pharmacokinetic Studies. Circulation. 2017 Sep 19;136(12):1102-1113. doi: 10.1161/CIRCULATIONAHA.117.028893. Epub 2017 Jul 20. PMID 28729250